CLINICAL TRIAL: NCT05253469
Title: Cryopreserved Aortic Homograft Versus Conventional Prosthetic Valves for Infective Endocarditis Involving the Aortic Valve : a Propensity Score Matched Analysis
Brief Title: Infective Endocarditis Surgery Using Conventional Prosthetic Valves Versus Cryopreserved Aortic Homograft
Acronym: IESCOPHO
Status: Enrolling by invitation | Type: Observational
Sponsor: Centre Cardiologique du Nord (Other)
Collaborators: Campus Bio-Medico University (Other); Henri Mondor University Hospital (Other); Universita degli Studi di Genova (Other); University of Bristol (Other); Aberdeen Royal Infirmary (Other)
Responsible Party: Sponsor
Other Study IDs: CN-21-24
Record Dates: First submitted 2022-02-14; First posted 2022-02-23 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Infective Endocarditis; Heart Failure
Keywords: IE ; CAH ; AVRpl ; Root replacement; Intervalvular fibrosa
MeSH Terms: conditions — Endocarditis; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cryopreserved Aortic Homograft: Include patients who received CAH for native (NVE) or prosthetic valve endocarditis (PVE).
  The CAH are implanted using miniroot procedure. For extended aortic valve infection, aortic root replacement and reconstruction of regional contiguity is the recommended approach. Complicated aortic IE may present with destruction of a large portion of the aortic annulus, annular abscess and colonization of infected foci in contiguous cardiac structures (eg. Aortic root and intervalvular fibrosa).
  Use of homograft in first time aortic valve replacement for IE decreased over time (9,4% to 5,6%) and in reoperation (37,5% to 28,5%) in a report from STS database between 2005-2011 (6). Nevertheless, the homograft was used more often in reoperations than in primary interventions (32.2% vs 7.0%, p < 0.0001) in both valve replacements (14,6%) and for root replacements (53,2%) (6).
  Interventions: Procedure: Cryopreserved Aortic Homograft; Procedure: Stented/Non stented xenograft; Procedure: Mechanical prostheses
- Stented/Non stented xenograft: Stented/Non stented xenograft may be inserted using separate or continuos stich with or without teflon pledget. The use of biological valves increased from 57% to 67% for primary the operation during which the use of mechanical valves decreased from 30% to 24%. For reoperations, the use of biologic valves increased from 38% to 52% compared to the warning use of mechanical valves from 20% to 17%. A homograft was used in only 2.5% of valve replacements, while a biological valve was used in 68.7% of the cases. This trend is reversed both in NVE and PVE the aortic root was involved (6). In the presence of peri-annular abscess formation and mitro-aortic discontinuity, conventional stented /non stented xenograft are used in combination with synthetic patch for both NVE and PVE.
  Interventions: Procedure: Cryopreserved Aortic Homograft; Procedure: Stented/Non stented xenograft; Procedure: Mechanical prostheses
- Mechanical valve prostheses: Mechanical prostheses may be inserted using separate or continuos stich with or without teflon pledget. Prior to 2000, mechanical valves were used in 50% of patients compared to 14% since 2009. Analysis of the STS Database (6) showed that from 2005 to 2011 a progressive shift in favour of biological valves both as the primary operation (NVE) (73%) and in the reoperation (PVE) (27%) compared to mechanical prosthesis. For extended aortic valve infection, aortic root replacement and reconstruction of regional contiguity is the recommended approach. Complicated aortic IE may present with destruction of a large portion of the aortic annulus, annular abscess and colonization of infected foci in contiguous cardiac structures (eg. aortic root and intervalvular fibrosa). In the presence of peri-annular abscess formation and mitro-aortic discontinuity, conventional mechanical prostheses are used in combination with synthetic patch for both NVE and PVE
  Interventions: Procedure: Cryopreserved Aortic Homograft; Procedure: Stented/Non stented xenograft; Procedure: Mechanical prostheses

INTERVENTIONS:
Procedure: Cryopreserved Aortic Homograft — CAH is used for aortic root reconstruction and for repair of mitro-aortic curtain (emicommando procedure) and it is inserted as miniroot . In cases of PVE the infected prosthesis is removed with aggressive debridement of all infected and necrotic tissue. (7)The coronary ostia are prepared for reconstruction of aortic root. In complex valve endocarditis involving aortic and mitral valve a double homograft may be used.Mitro-aortic endocarditis intervalvular fibrosa is largely involved.The abscess cavity is precisely bounded and debrided. and a double homograft is used for the reconstruction (commando procedure
  Other Names: Root replacement; Commando procedure; Emicommando procedure
Procedure: Stented/Non stented xenograft — The insertion of stented/non stented xenograft may be performed using separate or continuos stich with or without teflon pledget. Biological valves may be implated alone or combined with polyester or pericardial patch when reconstruction of annulus is required. In cases of aggressive lesions requiring root and /or intervalvular fibrosa reconstruction the choice of prosthetic bioroot using bioprosthetic valve is considered acceptable alternatives to CAH although it should be guided by the surgeon's experience
  Other Names: Root replacement; Commando procedure; Emicommando procedure
Procedure: Mechanical prostheses — The insertion of conventional mechanical valves may be performed using separate or continuos stich with or without teflon pledget. Mechanical prostheses may be implated alone or combined with polyester or pericardial patch when reconstruction of annulus is required. In cases of aggressive lesions requiring root and /or intervalvular fibrosa reconstruction the choice of prosthetic valved conduit with a mechanical valve is considered acceptable alternatives to CAH although it should be guided by the surgeon's experience
  Other Names: Root replacement; Commando procedure

SUMMARY:
: Evidence suggested that autologous or allogeneic tissue is more suitable to synthetic material in an infected field. Given the unwillingness of some surgeons to use artificial foreign materials, such as conventional mechanical or stent xenograft valve prostheses, cryopreserved aortic homografts (CAH) have been recommended revealing favorable outcomes in aortic valve endocarditis (AVE) surgery (1-5). This aspect is even more evident in cases involving prosthetic valve endocarditis (PVE) and other complex and aggressive lesions involving the aortic root and intervalvular fibrosa with abscess formation. However, most of these reports are fixed on single-arm observational studies without comparing CAH with conventional prostheses.

The key question of this study is to establish the difference in treatment failure (death, recurrent aortic valve regurgitation and reoperation), all-cause and cause-specific (cardiac vs noncardiac) mortality, hospitalizations for heart failure during follow-up (structural/non structural valve deterioration, thromboembolism and recurrent endocarditis) in patients who received the CAH vs conventional mechanical or stent xenograft valve prostheses for aortic valve replacement (AVR) secondary to infective endocarditis (IE)

DETAILED DESCRIPTION:
The target population enrolled in the study includes patients with aortic-valve endocarditis at risk of embolization, heart failure and uncontrolled infection undergoing AVR with the use of CAH or conventional mechanical or stent xenograft valve prostheses. Individuals were adequately treated per applicable standards, including for the treatment of infection, LV dysfunction and heart failure. Patients enrolled in the studies were NYHA functional class II, III, or outpatient NYHA IV.

Three groups of patients are included in the study. Patients who were managed with CAH, patients who received AVR with conventional stented xenograft and recipients of AVR undergoing surgery with the use of mechanical prostheses.

ELIGIBILITY:
Inclusion Criteria:

* Duke Criteria
* Uncontrolled Infection Local abscess Large vegetation False aneurysm, Fistula, Dehiscence of PV
* Embolism Large vegetation >10mm, persistent infection
* Heart Failure Involvement of aortic root, intervalvular fibrosa, pulmonary edema, cardiogenic shock

Exclusion Criteria :

* Pediatric
* Any echocardiographic evidence of absence of IE

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with aortic valve endocarditis with or without infection extending to other heart structures who were symptomatic of congestive heart failure and unresponsive to medical therapy and who were eligible for surgical aortic valve replacement. The severity of AMR was assessed by transthoracic echocardiography, performed using the European Society of Echocardiography criteria.
Sampling Method: Probability Sample
Enrollment: 760 (Estimated)
Dates: Start 2005-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | 10 years
  The primary end point of the study is the degree of treatment failure as assessed by death, recurrent aortic valve regurgitation and reoperation

SECONDARY OUTCOMES:
Overall Mortality | 10 years
  The secondary endpoint of the study is the evaluation of overall mortality
Cardiac Death | 10 years
  The secondary endpoint of the study is the evaluation of cardiac death
Non Cardiac Death | 10 years
  The secondary endpoint of the study is the evaluation of non cardiac death
Hospitalizations for Heart Failure (HF) | 10 years
  The secondary endpoint of the study is the evaluation of hospedalization rates for heart failure valve due to structural/non structural valve deterioration, thromboembolism and recurrent endocarditis
Major Adverse Cardiac or Cerebrovascular Events (MACCE) | 10 years
  Composite of major adverse cardiac or cerebrovascular events (rate of death, stroke, subsequent mitral valve surgery, hospitalization for heart failure, or an increase in New York Heart Association class higher than one), serious adverse events, recurrent aortic regurgitation, quality of life, and rehospitalization.
Echocardiographic Parameter Changes (LVEF) | 10 years
  Changes from baseline parameters including left ventricular ejection fraction
Echocardiographic Parameter Changes (recurrence) | 10 years
  Recurrent moderate-to-severe aortic regurgitation after intervention
Echocardiographic Parameter Changes (LVEDD) | 10 years
  Changes from baseline Left Ventricular End Diastolic Diameter
Echocardiographic Parameter Changes (Aortic Root diameter) | 10 years
  Changes from baseline aortic root diameter

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Nappi, MD, Principal Investigator — Centre Cardiologique du Nord
Locations (1):
- Francesco Nappi, Saint-Denis, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nappi F, Nenna A, Petitti T, Spadaccio C, Gambardella I, Lusini M, Chello M, Acar C. Long-term outcome of cryopreserved allograft for aortic valve replacement. J Thorac Cardiovasc Surg. 2018 Oct;156(4):1357-1365.e6. doi: 10.1016/j.jtcvs.2018.04.040. Epub 2018 Apr 18. PMID 29759737
- [Result] Olivito S, Lalande S, Nappi F, Hammoudi N, D'Alessandro C, Fouret P, Acar C. Structural deterioration of the cryopreserved mitral homograft valve. J Thorac Cardiovasc Surg. 2012 Aug;144(2):313-20, 320.e1. doi: 10.1016/j.jtcvs.2011.06.041. Epub 2011 Sep 8. PMID 21855094
- [Result] Nappi F, Spadaccio C, Dreyfus J, Attias D, Acar C, Bando K. Mitral endocarditis: A new management framework. J Thorac Cardiovasc Surg. 2018 Oct;156(4):1486-1495.e4. doi: 10.1016/j.jtcvs.2018.03.159. Epub 2018 Apr 13. No abstract available. PMID 29884490
- [Result] Nappi F, Spadaccio C, Acar C. Use of allogeneic tissue to treat infective valvular disease: Has everything been said? J Thorac Cardiovasc Surg. 2017 Apr;153(4):824-828. doi: 10.1016/j.jtcvs.2016.09.071. Epub 2016 Oct 24. No abstract available. PMID 27866779
- [Result] Kim JB, Ejiofor JI, Yammine M, Camuso JM, Walsh CW, Ando M, Melnitchouk SI, Rawn JD, Leacche M, MacGillivray TE, Cohn LH, Byrne JG, Sundt TM. Are homografts superior to conventional prosthetic valves in the setting of infective endocarditis involving the aortic valve? J Thorac Cardiovasc Surg. 2016 May;151(5):1239-46, 1248.e1-2. doi: 10.1016/j.jtcvs.2015.12.061. Epub 2016 Jan 23. PMID 26936004
- [Result] Sabik JF, Lytle BW, Blackstone EH, Marullo AG, Pettersson GB, Cosgrove DM. Aortic root replacement with cryopreserved allograft for prosthetic valve endocarditis. Ann Thorac Surg. 2002 Sep;74(3):650-9; discussion 659. doi: 10.1016/s0003-4975(02)03779-7. PMID 12238819
- [Result] Savage EB, Saha-Chaudhuri P, Asher CR, Brennan JM, Gammie JS. Outcomes and prosthesis choice for active aortic valve infective endocarditis: analysis of the Society of Thoracic Surgeons Adult Cardiac Surgery Database. Ann Thorac Surg. 2014 Sep;98(3):806-14. doi: 10.1016/j.athoracsur.2014.05.010. Epub 2014 Jul 29. PMID 25085561